CLINICAL TRIAL: NCT06436092
Title: Japanese Coronary Intervention Using Drug Eluting and Perfusion Therapy for Left Main Disease (JDEPTH-LM Registry)
Status: Recruiting | Type: Observational
Sponsor: TCROSS Co., Ltd. (Industry)
Collaborators: Kaneka Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: JDEPTH-LM Registry; jRCT1030240071 (Other: Japan Registry of Clinical Trials)
Record Dates: First submitted 2024-05-10; First posted 2024-05-30 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Stable Angina; Non-ST-elevation Acute Coronary Syndrome; Unstable Angina
Keywords: Ischemic heart disease
MeSH Terms: conditions — Angina, Stable; Angina, Unstable; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- JDEPTH-LM Registry Participants: Subjects ≥ 18 years of age with de novo LMD with LCx ostium stenosis presenting with stable angina, non-ST-elevation myocardial infarction, or unstable angina that are suitable for percutaneous coronary intervention including W-KBT processes. Approximately 280 subjects at 17 sites in Japan will be enrolled. Subjects will be followed through discharge and 12 months in routine clinical practice.

SUMMARY:
JDEPTH-LM Registry is a prospective, observational, multi-center study designed for the efficacy and safety of Double-effect kissing balloon technique (W-KBT) in left main (LM) bifurcation percutaneous coronary intervention (PCI) using Perfusion balloon (PB) and Drug coated balloon (DCB) in patients with left main coronary artery disease (LMD) with left circumflex artery (LCx) ostium stenosis.

DETAILED DESCRIPTION:
JDEPTH-LM Registry is a prospective observational multi-center study. The investigators will enroll and treat patients in the registry who meet the selection criteria under usual care and for whom PCI with W-KBT following on crossover stenting for LMT-LAD direction, proximal optimization technique (POT), and conventional kissing balloon technique (C-KBT) is the optimal treatment. The operators shall obtain oral or written consent from patients who meet the criteria before performing PCI, indicating the intention to perform PCI with W-KBT, and shall keep records. The investigators will continuously register cases attempting PCI with W-KBT according to the protocol and evaluate its efficacy and safety using data from this multi-center registry.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Patient with stable coronary artery disease, non-ST-elevation myocardial infarction, or unstable angina
3. Left main disease confirmed by coronary angiography or coronary CT angiography
4. Clinical and anatomical eligibility for PCI as agreed by the local Heart Team
5. Patient with consent prior to undergoing PCI
6. Left main Medina classification (1,1,1), (1,0,1), (0,1,1), (0,0,1) confirmed by coronary angiography
7. De novo target lesion in LMT-LAD amenable for crossover stenting with provisional side-branch approach as determined by PCI operator
8. De novo ostial LCx lesions
9. Lesion indicated in No. 8 with a length of less than 10 mm or a stenosis of less than 70% confirmed by coronary angiography

Exclusion Criteria:

1. Inability to provide written informed consent
2. Patient with a history of ST-elevation myocardial infarction within the previous 1 week
3. Patient in a state of cardiogenic shock
4. Patient with a history of coronary artery bypass grafting
5. Patient with malignant tumors or other conditions with a life expectancy of less than one year
6. Patient considered suitable for stent placement in the ostial LCx from a medical perspective
7. Patient considered unsuitable for anti-thrombotic therapy after PCI
8. Other patient whom the investigator deems unsuitable for the safe conduct of LM-PCI, including W-KBT

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects ≥ 18 years of age with de novo LMD with LCx ostium stenosis presenting with stable angina, non-ST-elevation myocardial infarction, or unstable angina that are suitable for percutaneous coronary intervention including W-KBT processes. Approximately 280 subjects at 17 sites in Japan will be enrolled. Subjects will be followed through discharge and 12 months in routine clinical practice.
Sampling Method: Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2024-05-27 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Procedure success rate | During PCI procedure
  indicating the proportion of cases meeting the following three conditions:
  * Device delivery success
  * Achievement of DCB expansion for 30 seconds or more
  * No bailout stenting performed in the LCx
Major adverse cardiovascular event (MACE) at 12 months | Within 12 months of PCI procedure
  consisting of all-cause mortality, nonfatal myocardial infarction (MI), and ischemia-driven unplanned revascularization for left main disease

SECONDARY OUTCOMES:
Time to ST-change from DCB inflation | During PCI procedure
  confirming the time from the initiation of W-KBT to any ST elevation/depression in the electrocardiogram (ECG) to evaluate the safety of the procedure
Total DCB Inflation time | During PCI procedure
  confirming the duration for which the inflation of the DCB can be sustained during W-KBT, as the recommendation time of DCB inflation is at least 30 seconds
Maximum changes in blood pressure and heart rate | During PCI procedure
  confirming the extent of blood pressure and heart rate changes resulting from maintaining W-KBT for 30 seconds or longer in the left main coronary trunk (LMT)
Rate of use of vasopressors, inotropes, and mechanical circulatory support systems after W-KBT | During PCI procedure
  confirming that hemodynamics is not disturbed by W-KBT for LMD
Incidence cases for each component of MACE and ischemia-driven unplanned revascularization for lesions at the LCx ostium | Within 12 months of PCI
  confirming the frequency of occurrences for each component of MACE

OTHER OUTCOMES:
Assessment of distal LAD coronary flow preservation during C-KBT vs. W-KBT | During PCI procedure
  Fractional flow reserve (FFR) values will be measured before and after each KBT, using either a conventional balloon or PB
ST-change recovery time | During PCI procedure
  confirming that ECG changes can easily recover even after W-KBT for LMD
Incidence of periprocedural MI defined by Fourth Universal Definition of Myocardial Infarction (4th UDMI), Academic Research Consortium (ARC)-2 and Society for Cardiovascular Angiography and Interventions (SCAI) definitions | Within 12 months of PCI
Incidence of LM stent deformation after W-KBT assessed by intravascular ultrasound (IVUS) | During PCI procedure
MACE at 12 months based on lesion characteristics at the LCx ostial lesions and the type of lesion preparation step | Within 12 months of PCI
Incidence of symptom onset during W-KBT and reviewing cases showing these symptoms | During PCI procedure
Incidence of Treatment Adverse Events [Safety and Tolerability] in patients with low left ventricular ejection fraction (LVEF) | During PCI procedure & Within 12 months of PCI
  The incidence rate will be calculated using the median LVEF or 40% as the cutoff
The procedural success rate based on the number of LM-PCI experiences | During PCI procedure & Within 12 months of PCI
  comparing efficacy and safety among various groups based on PCI operators' experience
Late lumen loss | During PCI procedure & Within 12 months of PCI
  in balloon dilated coverage area of the side branch lesion measured by QCA (Quantitative Coronary Angiography)
Assessment of ischemia including FFR or non-hyperemic pressure ratios (NHPRs) at follow-up visit | Within 12 months of PCI

CONTACTS AND LOCATIONS:
Locations (32):
- Japan (32):
  - Ichinomiya Municipal Hospital, Ichinomiya, Aichi-ken
  - Fujita Health University School of Medicine, Toyoake, Aichi-ken
  - Chiba University Hospital, Chiba, Chiba
  - New Tokyo Hospital, Matsudo, Chiba
  - Tokyo Bay Urayasu Ichikawa Medical Center, Urayasu, Chiba
  - Ehime Prefectural Central Hospital, Matsuyama, Ehime
  - Fukuoka Wajiro Hospital, Fukuoka, Fukuoka
  - National Hospital Organization Kyushu Medical Center, Fukuoka, Fukuoka
  - Kokura Memorial Hospital, Kitakyushu, Fukuoka
  - Gifu Heart Center, Gifu, Gifu
  - Gunma University Hospital, Maebashi, Gunma
  - Hakodate Municipal Hospital, Hakodate, Hokkaido
  - Sapporo Higashi Tokushukai Hospital, Sapporo, Hokkaido
  - Tsuchiura Kyodo General Hospital, Tsuchiura, Ibaraki
  - Tsukuba Medical Center Hospital, Tsukuba, Ibaraki
  - Kanazawa Cardiovascular Hospital, Kanazawa, Ishikawa-ken
  - Memorial Heart Center Iwate Medical University, Morioka, Iwate
  - Shonan Kamakura General Hospital, Kamakura, Kanagawa
  - Kitasato University School of Medicine, Sagamihara, Kanagawa
  - Yokosuka Kyosai Hospital, Yokosuka, Kanagawa
  - Chikamori Hospital, Kochi, Kochi
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - Shinshu University Hospital, Matsumoto, Nagano
  - Kurashiki Central Hospital, Kurashiki, Okayama-ken
  - Urasoe General Hospital, Urasoe, Okinawa
  - The University of Tokyo Hospital, Bunkyo, Tokyo
  - Moriyama Memorial Hospital, Edogawa City, Tokyo
  - Sakakibara Heart Institute, Fuchū, Tokyo
  - Jikei University Katsushika Medical Center, Katsushika-ku, Tokyo
  - NTT Medical Center Tokyo, Shinagawa, Tokyo
  - Keio University Hospital, Shinjuku, Tokyo
  - Japanese Red Cross Wakayama Medical Center, Wakayama, Wakayama

IPD SHARING:
Plan to Share IPD: No